CLINICAL TRIAL: NCT02928380
Title: A Clinical Study to Evaluate the Ability of an Experimental Denture Adhesive to Prevent Food Particle Ingress Under Dentures
Brief Title: Evaluation of a Experimental Denture Adhesive to Prevent Food Ingress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 205915
Record Dates: First submitted 2016-07-18; First posted 2016-10-10 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-07

CONDITIONS: Denture Retention

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Reference Denture Adhesive (Active Comparator): Participants applied reference denture adhesive as a 3 dabs those were applied to upper denture and 2 dabs those were applied to lower denture which were placed in the mouth.
  Interventions: Device: Reference (Marketed) Denture Adhesive
- Test Denture Adhesive (Experimental): Participants applied test denture adhesive as 3 continuous strips those were applied to upper denture and one continuous strip that was applied to the lower denture, which were placed in the mouth.
  Interventions: Device: Experimental Denture Adhesive
- No Adhesive (Negative Control) (No Intervention): Participants did not apply any denture adhesive in this treatment arm.

INTERVENTIONS:
Device: Experimental Denture Adhesive — Participants received a single application of test denture adhesive with a Flat Ribbon Nozzle as 3 Continuous strips those were applied to upper denture and one continuous strip that was applied to the lower denture which were placed in the mouth.
  Arms: Test Denture Adhesive
Device: Reference (Marketed) Denture Adhesive — Participants received a single application of marketed denture adhesive with a flat ribbon nozzle as a 3 dabs those were applied to upper denture and 2 dabs those were applied to lower denture, which were placed in the mouth.
  Arms: Reference Denture Adhesive

SUMMARY:
In this clinical study, an experimental denture adhesive with a precision tip nozzle was tested to evaluate the relative efficacy to reduce the ingress of food under the denture compared to use of no adhesive or a standard marketed adhesive.

DETAILED DESCRIPTION:
The aim of this study is to explore the mass of food particle ingress when an adhesive is extruded through the new nozzle with directed application compared to the use of no adhesive and a marketed adhesive (extruded through a flat ribbon nozzle [FRN]) with standard application as per product label, utilizing a peanut occlusion methodology. This was a single center, controlled, single blind (to the examiner performing the safety assessments (oral soft tissue [OST] examination) and the laboratory staff weighing the peanut particles), randomized, three-treatment, three-period, cross-over design in participants with full upper and lower dentures. Each treatment period consisted of one day of testing with at least two days between treatment visits. This study consisted four visits: Visit 1 - Screening Visit; Visit 2 - Treatment 1 Visit; Visit 3 - Treatment 2 Visit and Visit 4 - Treatment 3 Visit.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Aged between 18 and 85 years inclusive
* Understands and is willing, able and likely to comply with all study procedures and restrictions
* Good general and mental health with, in the opinion of the investigator or medically qualified designee:No clinically significant and relevant abnormalities of medical or physical history; Absence of any condition that would impact on the participant's safety or well being or affect the individual's ability to understand and follow study procedures
* A qualifying full denture in both the upper and lower arch
* Dentures are well fitting (Kapur (Olshan Modification) Retention and Stability Index Sum Score ≥6)
* Dentures are well made (according to the well-made assessment)
* Participants must report that they get food trapped under their denture
* A peanut particle migration rating >0 for both dentures at screening

Exclusion Criteria:

* Women who are known to be pregnant (participant-reported) or who are intending to become pregnant over the duration of the study
* Women who are breast-feeding
* Medications, which in the opinion of the investigator, would interfere with the conduct of the study
* Taking or have taken a bisphosphonate drug for treatment of osteoporosis
* A serious chronic disease requiring hospitalization
* History of swallowing difficulties or choking
* Any condition not previously mentioned that in the investigator's opinion may impair the study evaluation
* Any condition or medication which, in the opinion of the investigator, is currently causing xerostomia
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients
* Known allergy to peanuts or any other nut
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit
* Previous participation in this study
* Recent history (within the last year) of alcohol or other substance abuse
* OST examination findings such as stomatitis, open sores, lesions, redness or swelling
* An employee of the sponsor or the study site or members of their immediate family
* Any participant who, in the opinion of the Investigator, should not participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2016-07-25 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fort Wayne, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single center in the United States.
Pre-assignment Details: A total of 91 participants were screened, out of which only 83 participants were randomized to the study. 8 participants were not randomized: 7 participants due to screening failure and 1 participant due lost to follow up.
Groups:
- Reference Denture Adhesive/Test Denture Adhesive/No Adhesive: Participants received reference denture adhesive, test denture adhesive and no adhesive by site staff in treatment periods 1, 2, 3 respectively, to their dentures which were placed in their mouth. A single application of each adhesive was applied. The three treatment periods were separated by a washout period of 2-7 days.
- Reference Denture Adhesive/No Adhesive/Test Denture Adhesive: Participants received reference denture adhesive, no adhesive and test denture adhesive by site staff in treatment periods 1, 2, 3 respectively, to their dentures which were placed in their mouth. A single application of each adhesive was applied. The three treatment periods were separated by a washout period of 2-7 days.
- Test Denture Adhesive/Reference Denture Adhesive/No Adhesive: Participants received test denture adhesive, reference denture adhesive and no adhesive by site staff in treatment periods 1, 2, 3 respectively, to their dentures which were placed in their mouth. A single application of each adhesive was applied. The three treatment periods were separated by a washout period of 2-7 days.
- Test Denture Adhesive/No Adhesive/Reference Denture Adhesive: Participants received test denture adhesive, no adhesive and reference denture adhesive by site staff in treatment periods 1, 2, 3 respectively, to their dentures which were placed in their mouth. A single application of each adhesive was applied. The three treatment periods were separated by a washout period of 2-7 days.
- No Adhesive/Reference Denture Adhesive/Test Denture Adhesive: Participants received no adhesive, reference denture adhesive and test denture adhesive by site staff in treatment periods 1, 2, 3 respectively, to their dentures which were placed in their mouth. A single application of each adhesive was applied. The three treatment periods were separated by a washout period of 2-7 days.
- No Adhesive/Test Denture Adhesive/Reference Denture Adhesive: Participants received no adhesive, test denture adhesive and reference denture adhesive by site staff in treatment periods 1, 2, 3 respectively, to their dentures which were placed in their mouth. A single application of each adhesive was applied. The three treatment periods were separated by a washout period of 2-7 days.
Period: Period 1
Arm/Group | Reference Denture Adhesive/Test Denture Adhesive/No Adhesive | Reference Denture Adhesive/No Adhesive/Test Denture Adhesive | Test Denture Adhesive/Reference Denture Adhesive/No Adhesive | Test Denture Adhesive/No Adhesive/Reference Denture Adhesive | No Adhesive/Reference Denture Adhesive/Test Denture Adhesive | No Adhesive/Test Denture Adhesive/Reference Denture Adhesive
Started | 13 | 14 | 14 | 14 | 14 | 14
Completed | 13 | 14 | 14 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Wash Out Period 1
Arm/Group | Reference Denture Adhesive/Test Denture Adhesive/No Adhesive | Reference Denture Adhesive/No Adhesive/Test Denture Adhesive | Test Denture Adhesive/Reference Denture Adhesive/No Adhesive | Test Denture Adhesive/No Adhesive/Reference Denture Adhesive | No Adhesive/Reference Denture Adhesive/Test Denture Adhesive | No Adhesive/Test Denture Adhesive/Reference Denture Adhesive
Started | 13 | 14 | 14 | 14 | 14 | 14
Completed | 13 | 14 | 14 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Reference Denture Adhesive/Test Denture Adhesive/No Adhesive | Reference Denture Adhesive/No Adhesive/Test Denture Adhesive | Test Denture Adhesive/Reference Denture Adhesive/No Adhesive | Test Denture Adhesive/No Adhesive/Reference Denture Adhesive | No Adhesive/Reference Denture Adhesive/Test Denture Adhesive | No Adhesive/Test Denture Adhesive/Reference Denture Adhesive
Started | 13 | 14 | 14 | 14 | 14 | 14
Completed | 13 | 14 | 14 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Wash Out Period 2
Arm/Group | Reference Denture Adhesive/Test Denture Adhesive/No Adhesive | Reference Denture Adhesive/No Adhesive/Test Denture Adhesive | Test Denture Adhesive/Reference Denture Adhesive/No Adhesive | Test Denture Adhesive/No Adhesive/Reference Denture Adhesive | No Adhesive/Reference Denture Adhesive/Test Denture Adhesive | No Adhesive/Test Denture Adhesive/Reference Denture Adhesive
Started | 13 | 14 | 14 | 14 | 14 | 14
Completed | 13 | 14 | 14 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Reference Denture Adhesive/Test Denture Adhesive/No Adhesive | Reference Denture Adhesive/No Adhesive/Test Denture Adhesive | Test Denture Adhesive/Reference Denture Adhesive/No Adhesive | Test Denture Adhesive/No Adhesive/Reference Denture Adhesive | No Adhesive/Reference Denture Adhesive/Test Denture Adhesive | No Adhesive/Test Denture Adhesive/Reference Denture Adhesive
Started | 13 | 14 | 14 | 14 | 14 | 14
Completed | 13 | 14 | 14 | 14 | 14 | 14
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis was performed on Intention to treat (ITT) population which included all participants who were randomized, received at least one dose of study treatment and had at least one post baseline efficacy assessment.
Groups:
- Overall Participants: All the participants received all three treatments (reference denture adhesive, test denture adhesive and no adhesive) in the study period 1, 2, and 3 according to the randomization sequence. Each treatment period was separated by washout period of 2-7 days. All randomized participants were included for baseline evaluation.
Arm/Group | Overall Participants
Number analyzed (Participants) | 83
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (12.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 82
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 12
  White | 70
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Combined Mass of Peanuts (Gram) (From Upper and Lower Dentures) for Reference Denture Adhesive and on no Adhesive Use
Description: Participants were provided with 30-32 g (accurately weighed) non-salted peanuts, divided into smaller portions of approximately four whole peanuts. Each portion chewed for approximately 20 seconds. After completion of the peanut consumption, participants rinsed their mouth with water, participants may remove any residual peanut particles from their mouth with water and a gauze pad. Participants than removed their dentures. Peanut particles were collected from the fit surfaces of the dentures and the gauzes, and weighed to evaluate the mass of food particles that had migrated under the denture (keeping the particles associated with the upper and lower dentures separate).
Time Frame: Up to 17 days
Population: Analysis for this outcome was performed on ITT population including all participants who were randomized, received at least one dose of study treatment and had at least one post baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: gram (g)
Groups:
- Reference Denture Adhesive: Participants received reference denture adhesive by site staff as a 3 dabs those were applied to upper denture and 2 dabs those were applied to lower denture which were placed in the mouth.
- No Adhesive (Negative Control): Participants did not receive any denture adhesive by site staff in this treatment arm.
Arm/Group | Reference Denture Adhesive | No Adhesive (Negative Control)
Number analyzed (Participants) | 83 | 83
gram (g) | 0.06 (0.057) | 0.08 (0.151)
Statistical Analysis 1: Comparison: Reference Denture Adhesive vs No Adhesive (Negative Control); H0: The mean mass of food particles retrieved from using a marketed denture adhesive with a flat ribbon nozzle is no different from using no adhesive H01: The mean mass of food particles retrieved from using a marketed denture adhesive with a flat ribbon nozzle is different from using no adhesive; Test type: Other; p = 0.0987, ANOVA; ANOVA Model with weight of the peanut particle (food occlusion) as response variable, treatment and period as fixed effect; Least square (LS) mean difference = -0.02, 95% CI 2-sided [-0.05 to 0.00] — Difference is first named treatment minus second named treatment is such that a negative difference favors the first named treatment

2. Secondary Outcome: Combined Mass of Peanuts (Gram) (From Upper and Lower Dentures) for an Experimental Denture Adhesive and on no Adhesive Use
Description: as for outcome 1
Time Frame: Up to 17 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g
Groups:
- Test Denture Adhesive: Participants received test denture adhesive by site staff as 3 continuous strips those were applied to upper denture and one continuous strip that was applied to the lower denture, which were placed in the mouth.
Arm/Group | Test Denture Adhesive | No Adhesive (Negative Control)
Number analyzed (Participants) | 83 | 83
g | 0.07 (0.092) | 0.08 (0.151)

3. Secondary Outcome: Combined Mass of Peanuts (Gram) (From Upper and Lower Dentures) for an Experimental Denture Adhesive and Reference Denture Adhesive
Description: as for outcome 1
Time Frame: up to 17 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Test Denture Adhesive | Reference Denture Adhesive
Number analyzed (Participants) | 83 | 83
g | 0.07 (0.092) | 0.06 (0.057)

4. Secondary Outcome: Composite Kapur (Olshan Modification) Index Scores for Denture Retention and Stability
Description: Kapur (Olshan modification) Index score was assessed to examine each denture (upper & lower) for retention & stability. Retention was measured as score of 0-5 to assess nature of resistance offered by denture to vertical pull & lateral force: 5=Excellent;4=Very Good;3=Good;2=Fair;1= Poor;0=No retention. Stability was measured as score of 0-4 to assess nature of rocking offered by denture base on its supporting structures under pressure:4=Excellent (no rocking);3=Good (very slight rocking);2=Fair (slight rocking);1=Poor (moderate rocking);0=No stability (extreme rocking). Composite Kapur (Olshan modification) Index scores was measured as the sum score of retention & stability for upper or lower dentures separately such that a sum score of zero represents no retention and stability and a sum score of 9 represents excellent retention and stability.
Time Frame: Up to 17 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Reference Denture Adhesive | Test Denture Adhesive | No Adhesive (Negative Control)
Number analyzed (Participants) | 83 | 83 | 83
scores on a scale
  For Upper Denture | 8.67 (0.828) | 8.84 (0.594) | 8.35 (1.224)
  For Lower Denture | 7.42 (1.815) | 8.11 (1.593) | 6.36 (1.535)

5. Secondary Outcome: Kapur (Olshan Modification) Index Scores for Denture Retention
Description: Kapur (Olshan modification) Index scores were assessed to examine each denture (upper & lower) for its retention ability. Retention was measured as score of 0-5 to assess nature of resistance offered by denture to vertical pull & lateral force: 5=Excellent - denture offered excellent resistance to vertical pull and lateral force; 4= Very Good- denture offered very good resistance to vertical pull and lateral force; 3= Good- denture offered moderate resistance to vertical pull and lateral force; 2= Fair- denture offered moderate resistance to vertical pull and little or no resistance to lateral forces; 1= Poor- denture offers slight resistance to vertical pull and little or no resistance to lateral force; 0= No retention- when the denture was seated in place, it displaced itself. Higher the score, higher the retention ability of denture.
Time Frame: Up to 17 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Reference Denture Adhesive | Test Denture Adhesive | No Adhesive (Negative Control)
Number analyzed (Participants) | 83 | 83 | 83
scores on a scale
  For Upper Denture | 4.80 (0.512) | 4.90 (0.335) | 4.63 (0.728)
  For Lower Denture | 4.05 (1.070) | 4.43 (0.940) | 3.46 (0.874)

6. Secondary Outcome: Kapur (Olshan Modification) Index Scores for Denture Stability
Description: Kapur (Olshan modification) Index scores were assessed to examine each denture (upper & lower) for its stability ability. Stability was measured using score of 0-4: 4= Excellent- when denture base offered no rocking on its supporting structures under pressure; 3= Good- when denture base had very slight rocking on its supporting structures under pressure; 2= Fair- when denture base had slight rocking on its supporting structures under pressure; 1= Poor- when denture base had moderate rocking on its supporting structures under pressure; 0= No stability- when denture base had extreme rocking under pressure. Higher the score, higher the stability ability of denture.
Time Frame: Up to 17 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Reference Denture Adhesive | Test Denture Adhesive | No Adhesive (Negative Control)
Number analyzed (Participants) | 83 | 83 | 83
scores on a scale
  For Upper Denture | 3.88 (0.363) | 3.94 (0.286) | 3.72 (0.570)
  For Lower Denture | 3.37 (0.807) | 3.67 (0.700) | 2.90 (0.775)

ADVERSE EVENTS:
Arm/Group | Reference Denture Adhesive | Test Denture Adhesive | No Adhesive (Negative Control)
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/83 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/83 | 0/83
Other Adverse Events (participants affected / at risk) | 0/83 | 0/83 | 0/83

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.